CLINICAL TRIAL: NCT00097617
Title: National Cooperative Growth Study (NCGS) of Nutropin AQ, Nutropin, and Protropin in Children With Growth Failure Due to Chronic Renal Insufficiency (CRI) or End Stage Renal Disease (ESRD)
Brief Title: A Study in Children With Growth Failure Due to Chronic Renal Insufficiency (CRI) or End Stage Renal Disease (ESRD)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 85-036, Substudy 11
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Renal Insufficiency; End-Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is a multicenter, open-label, observational, postmarketing surveillance study that will collect information on the use of Genentech growth hormone (GH) preparations to treat children with CRI in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with CRI or ESRD and treated with a Genentech GH preparation on or after 1 January 2001
* CRI documented using the Schwartz formula indicates a calculated creatinine clearance (CrCl) of <=75 mL/min/1.73 m^2
* Ability to keep follow up appointments throughout the study

Exclusion Criteria:

* Subjects receiving a non-Genentech GH preparation
* Subjects with closed epiphyses
* Subjects with active neoplasia
* Current participation in another GH clinical study
* Current participation in the core study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2002-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lippe, M.D., Study Director — Genentech, Inc.